CLINICAL TRIAL: NCT02351076
Title: Correlation of Right-left Shunt Detection in Cardioembolism Etiology in Stroke Patient. Pilot Study.
Brief Title: Correlation of Right-left Shunt Detection in Cardioembolism Etiology in Stroke Patient.
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: RVO-FNOs/2014
Record Dates: First submitted 2014-11-23; First posted 2015-01-30 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Foramen Ovale Patent
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to compare correlation for right to left shunts (mainly patent foramen ovale) detection for three methods-transesophageal echo as a gold standard, transcranial doppler with contrast agent (microbubbles) and new method- Flow detection system ( Cardiox TM) in young stoke patients ( age under 55 years).

DETAILED DESCRIPTION:
The aim of the study is to compare correlation for right to left shunts (mainly patent foramen ovale) detection for three methods-transesophageal echo as a gold standard, transcranial doppler with contrast agent (microbubbles) and new method- Flow detection system ( Cardiox TM) in young stoke patients ( age under 55 years). Flow detection systém is a new method for right to left shunt detection comfortable for patients, not dependent on experienced examinator and only one method with exact valsalve maneuver measurement. Right to left shunt could be important etiology of cardioembolization in young stroke patient population, therefore screening for this condition is recommended in all young patient after ischemic stroke especially with unclear etiology. Flow detection systes seams to be ideal screening method for this patients.

ELIGIBILITY:
Inclusion Criteria:ischemic stroke / TIA, signed informed consent -

Exclusion Criteria:imposibillity to undergo transesophageal echo, transcranial doppler with contrast or Cardiox flow detection system

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient after ischemic stroke including TIA, age 18-55 year
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
detection of right-to-left shunt | 1 week
  Correletation of right-to-left shunt detection by 3 methods: transesophageal echocardiography, transcranial Doppler with contrast agent (microbubbles) and Flow detection system (Cardiox TM)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kuliha, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No